CLINICAL TRIAL: NCT03905057
Title: Effect of Early Shockwave Therapy Protocol for Preservation and Restoration of Erectile Function After Nerve-sparing Radical Prostatectomy
Brief Title: Early Shockwave Therapy for Post-RP ED
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dornier MedTech Systems (Industry)
Collaborators: Hospital Universitari de Bellvitge (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EspPRP-ED_001
Record Dates: First submitted 2019-03-26; First posted 2019-04-05 (Actual); Last update posted 2019-04-08 (Actual); Status verified 2019-04

CONDITIONS: Erectile Dysfunction Following Radical Prostatectomy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sham ESWT + 5mg Tadalafil (Sham Comparator): Patients will receive shockwave treatments (12 sessions for all subjects, 5000 shockwaves at each session), using a sham applicator which is highly similar to the active applicator except that the sham applicator does not emit shockwaves, twice a week (total of 6 weeks) without treatment interval. Patients will receive Tadalafil 5mg for 24 weeks daily beginning the day of removal of the urinary catheter.
  Interventions: Device: Dornier Aries 2 (with sham applicator)
- Active ESWT + 5mg Tadalafil (Active Comparator): Patients will receive shockwave treatments (12 sessions for all subjects, 5000 shockwaves at each session), twice a week (total of 6 weeks). Patients will receive Tadalafil 5mg for 24 weeks daily beginning the day of removal of the urinary catheter.
  Interventions: Device: Dornier Aries 2 (with active applicator)

INTERVENTIONS:
Device: Dornier Aries 2 (with active applicator) — Active ESWT: 5000 shockwaves per session. 2 ESWT sessions per week, 12 sessions in total.
  Arms: Active ESWT + 5mg Tadalafil
Device: Dornier Aries 2 (with sham applicator) — Sham ESWT - No shockwave administered
  Arms: Sham ESWT + 5mg Tadalafil

SUMMARY:
This pilot study aims to explore the feasibility, safety and effectiveness of two different extracorporeal shock wave therapy (ESWT) protocols for patients receiving nerve-sparing radical prostatectomy (RP).

DETAILED DESCRIPTION:
This is an open-label, randomized, 2-parallel-arm trial (n=94). All patients will receive (A) sham (n=47) or (B) active ESWT (n=47) twice/week for 6 weeks (12 sessions total). Concurrently, all patients will receive daily tadalafil 5mg for 24 weeks. Patients will then undergo a 4 week washout period without erectogenic aids, and return for a 28-week evaluation. Subsequently, patients requiring further erectogenic aids after 28 weeks will be offered intracavernosal injections (ICI) of prostaglandin E1 (PGE1).

Random assignment will be performed by computer program (eg. randomizer.org), in a design that obtains equal sample size per group.

All patients will be followed for a period of 24 months post-RP. Follow-up protocol includes evaluation of the IIEF, EHS, GAQ, ICI usage and tolerability, stretched flaccid penile length, urinary incontinence, and oncologic status.

ELIGIBILITY:
Inclusion Criteria:

* Men scheduled for robotic bilateral nerve-sparing radical prostatectomy
* Diagnosed with low/intermediate-risk prostate cancer:

  * PSA < 20 ng/ml
  * Gleason score < 8
  * PCa stage =< T2b
* Baseline IIEF-ED 22-30 without erectogenic aids
* No urinary incontinence (no usage of urinary pads)
* Sexually active, in a stable heterosexual relationship
* Able to understand and complete patient questionnaires
* Consent to participate

Exclusion Criteria:

* Anatomical abnormalities in the genitalia or pelvic region
* Post-RP complications that could impact safety or effectiveness of ESWT (eg. hematoma, fistula, unresolved anastomotic leak)
* Incomplete tumor removal (positive surgical margin)
* Tumor upstaging beyond T2b
* Nerve sparing score < 4
* Previous or scheduled treatment with pelvic radiotherapy and/or androgen deprivation therapy
* Untreated hypogonadism (serum total testosterone < 300 mg/dL)
* Anti-coagulant medication, or any blood coagulation disorders (INR > 3)
* Any other condition that would prevent the patient from completing the study, as judged by the principle investigator

Ages: 50 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2018-03-26 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
The difference in average Erectile Function (EF) domain score of the International Index of Erectile Function (IIEF) between the groups at 28-week follow up | 28-week follow up visit
  EF domain of the IIEF questionnaire will be completed. IIEF-EF consists of items 1,2,3,4,5,15 of the IIEF questionnaire.According to the score of the iIEF-EF there are five categories of erectile function: 1-10 (Severe Erectile Dysfunction), 11-16(Moderate dysfunction), 17-21(Mild to moderate dysfunction), 22-25(Mild dysfunction), 26-30 (No dysfunction)
The difference in average Erectile Function (EF) domain score of the International Index of Erectile Function (IIEF) between the groups at 24-month follow up | 24-month follow up visit
  EF domain of the IIEF questionnaire will be completed. IIEF-EF consists of items 1,2,3,4,5,15 of the IIEF questionnaire.According to the score of the iIEF-EF there are five categories of erectile function: 1-10 (Severe Erectile Dysfunction), 11-16(Moderate dysfunction), 17-21(Mild to moderate dysfunction), 22-25(Mild dysfunction), 26-30 (No dysfunction)

SECONDARY OUTCOMES:
Proportion of patients achieving Erectile Function (EF) domain score of the International Index of Erectile Function (IIEF) of 22-30 in each group | baseline, 12-weeks post-RP, 24-weeks post-RP, 28-weeks post-RP, 52-weeks post-RP, 18-months post-RP and 24-months post-RP
  The proportion of patients achieving Erectile Function (EF) domain score of the International Index of Erectile Function (IIEF) of 22-30 (indicating mild to no erectile dysfunction) in each group. EF domain of the IIEF questionnaire will be completed. IIEF-EF consists of items 1,2,3,4,5,15 of the IIEF questionnaire.According to the score of the iIEF-EF there are five categories of erectile function: 1-10 (Severe Erectile Dysfunction), 11-16(Moderate dysfunction), 17-21(Mild to moderate dysfunction), 22-25(Mild dysfunction), 26-30 (No dysfunction).
Change in each domain of the full International Index of Erectile Function (IIEF) score | baseline, 12-weeks post-RP, 24-weeks post-RP, 28-weeks post-RP, 52-weeks post-RP, 18-months post-RP and 24-months post-RP
  Change in each domain of the full International Index of Erectile Function (IIEF) score from baseline and from each follow-up. EF domain of the IIEF questionnaire will be completed. IIEF-EF consists of items 1,2,3,4,5,15 of the IIEF questionnaire.According to the score of the iIEF-EF there are five categories of erectile function: 1-10 (Severe Erectile Dysfunction), 11-16(Moderate dysfunction), 17-21(Mild to moderate dysfunction), 22-25(Mild dysfunction), 26-30 (No dysfunction)
Change in Erection Hardness Score | baseline, 12-weeks post-RP, 24-weeks post-RP, 28-weeks post-RP, in-office ICI visits, 52-weeks post-RP, 18-months post-RP and 24-months post-RP
  The Erection Hardness Score (EHS) is a single-item Likert scale to assess erectile dysfunction. Male patients have to answer the question "How would you rate the hardness of your erection?". They answer by selecting from the following options: 0 = Penis does not enlarge; 1 = Penis is large, but not hard; 2 = Penis is hard, but not hard enough for penetration; 3 = Penis is hard enough for penetration, but not completely hard; 4 = Penis is completely hard and fully rigid.
Change in Global Assessment Questionnaire (GAQ) score | 12-weeks post-RP, 24-weeks post-RP, 28-weeks post-RP, 52-weeks post-RP, 18-months post-RP and 24-months post-RP
  The Global Assessment Questionnaire (GAQ) is a tool to evaluate the efficacy of the treatment. Patients will be asked and provide scores (on a scale of 1 to 5) for treatment related, with a score of 1 being least favourable and 5 being most favourable.
Change in stretched flaccid penile length | baseline, 12-weeks post-RP, 24-weeks post-RP, 52-weeks post-RP, 18-months post-RP and 24-months post-RP
  The flaccid penis of each patient will be stretched and measured from the base of the penis to the tip of the glans.
Change in degree of incontinence | First treatment session, 12-weeks post-RP, 24-weeks post-RP, 52-weeks post-RP, 18-months post-RP and 24-months post-RP
  Incontinence will be determined by the number of pads used per day and the time to achieve 0-1 pad will be compared between the groups.
Oncologic status | 12-weeks post-RP, 24-weeks post-RP, 52-weeks post-RP, 18-months post-RP and 24-months post-RP
  The oncologic status of each patient will be evaluated determined by the serum prostate specific antigen (PSA) levels.
Time to recovery of penetration erection hardness without erectogenic aids | baseline, 12-weeks post-RP, 24-weeks post-RP, 28-weeks post-RP, in-office ICI visits, 52-weeks post-RP, 18-months post-RP and 24-months post-RP
  Penetration erection hardness is having an EHS score of 3-4. The Erection Hardness Score (EHS) is a single-item Likert scale to assess erectile dysfunction. Male patients have to answer the question "How would you rate the hardness of your erection?". They answer by selecting from the following options: 0 = Penis does not enlarge; 1 = Penis is large, but not hard; 2 = Penis is hard, but not hard enough for penetration; 3 = Penis is hard enough for penetration, but not completely hard; 4 = Penis is completely hard and fully rigid.
Tolerability to and reliance on intracavernosal injections for satisfactory erections: Visual Analog Scale for Pain | ICI visits, 52-weeks post-RP, 18-months post-RP and 24-months post-RP
  Patients who are unsatisfied with their erectile function at the 28 week visit, will be offered intracavernosal injections (10mg PGE1, 2x/week) for the remaining duration of the study. During each in-office ICI, patients will report pain tolerability (Visual Analog Scale for Pain), and maximum EHS achieved. Patients will be allowed to stop ICI if they report satisfactory erections without any erectogenic aids for 2 weeks. Patients will be allowed to resume ICI if erectile function decreases, and they report unsatisfactory erections with erectogenic aids for 2 weeks. Dates of stopping and/or resuming ICI will be recorded. At the 52 weeks, 18 and 24 months post-RP follow-up sessions, All patients will self-administer ICI of 10mg PGE1 during the visit, and report pain tolerability (Visual Analog Scale for Pain), and maximum EHS achieved.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona, Spain